CLINICAL TRIAL: NCT01437371
Title: Is There a Benefit to Optimize HF (Heart Failure) Treatment in Aged Over 80 Year's Old Patients?
Brief Title: Is There a Benefit to Optimize Heart Failure (HF) Treatment in Aged Over 80 Year's Old Patients?
Acronym: HF 80
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Servier (Industry); LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0102
Record Dates: First submitted 2011-08-31; First posted 2011-09-20 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
Keywords: Heart failure; Aged and over 80; clinical trial; quality of life
MeSH Terms: conditions — Heart Failure | interventions — Captopril; Lisinopril; Ramipril; trandolapril

ARMS (2):
- optimized (Other): The purpose of this study is to determine if there is an interest to optimize HF management in patients over 80 years old. The primary objective is to assess the effect of HF optimized management (guidelines of the European society of Cardiology (ESC) on QOL in aged over 80 year's old at 6 months
  Interventions: Drug: - Angiotensin conversing enzyme inhibitors: enalapril, captopril, lisinopril, ramipril, trandolapril.
- usual care (Other)
  Interventions: Drug: - Angiotensin conversing enzyme inhibitors: enalapril, captopril, lisinopril, ramipril, trandolapril.

INTERVENTIONS:
Drug: - Angiotensin conversing enzyme inhibitors: enalapril, captopril, lisinopril, ramipril, trandolapril. — The purpose of this study is to determine if there is an interest to optimize HF management in patients over 80 years old. The primary objective is to assess the effect of HF optimized management (guidelines of the European society of Cardiology (ESC) on QOL in aged over 80 year's old at 6 months

SUMMARY:
The purpose of this study is to determine if there is an interest to optimize HF (heart failure) management in patients over 80 years old. The primary objective is to assess the effect of HF (heart failure) optimized management (guidelines of the European society of Cardiology (ESC) on Quality of Life (QOL) in aged over 80 year's old at 6 months.

DETAILED DESCRIPTION:
Aging population, and better management of various heart diseases including ischemic explain the growing up of incidence and prevalence of chronic heart failure. The aging of the population leads now to support services in cardiology and particularly in the units of heart failure in subjects over 80 years. It's a special population with several co-morbidities, in whom it is difficult to introduce all the recommended treatments with optimal doses. There is indeed a significant difference between the optimal doses of treatments tested in studies on heart failure and doses found on the orders of inpatients for HF (heart failure). Unfortunately clinical trials on heart failure have recruited young patients, mean age 65 years. Clinical studies in cardiology and particularly in heart failure recruit young subjects at the expense of seniors who are underrepresented in these studies.

The investigators will compare two groups: the first one with an "optimized" management and the second one as "usual care".

The primary endpoint will evaluate the quality of life at 6 months according to the scale of Minnesota. Secondary outcomes will be the quality of life at 12 months, quality of life measured by the SF 12 (to check what level is most suited to this population) at baseline, 6 months and one year, mortality at 12 months, the number of re-hospitalization and cardiovascular events at 12 months, New York Health Association (NYHA) class (at baseline, 6 months and 12 months) and walking test for 6 minutes (at baseline, 6 months and 12 months). Finally the investigators plan to conduct an analysis on the medical and economic interest of this support.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 80 year's old subjects
* Hospitalized for an acute heart failure
* Left Ventricle Ejection Fraction ≤ 35%
* Evaluated life expectancy (Seattle HF score) > 1 year

Exclusion Criteria:

* Dementia
* Does not understand French language
* Followed with an optimized management
* With reduced mobility
* Recruited in another clinical trial or in a HF management network
* AHF with curable aetiology : cardiovascular surgery for CABG or valvular replacement, angioplasty
* MDRD < 30 ml/min/1.73m²

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of life | baseline, at 6 months

SECONDARY OUTCOMES:
Mortality | at 12 months
Rehospitalisation | at 12 months
Cardiovascular events | at 12 months
Cardiac fibrosis | at 12 months
Quality of life | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain ESCHALIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Eschalier R, Jean F, Pereira B, Monzy S, Vorilhon C, Mactoux V, Citron B, Sapin V, Motreff P, Lusson JR. Is there benefit in optimising heart failure treatment in over-80 year-old patients? (HF-80 study): study protocol for a randomized controlled trial. Trials. 2012 Mar 6;13:25. doi: 10.1186/1745-6215-13-25. PMID 22394464